CLINICAL TRIAL: NCT01565135
Title: Immunization Delivery in Obstetrics and Gynecology Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11-1149; U01IP000501 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Immunization Status Among Obstetrics and Gynecology Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Practices (Experimental): Intervention offices will adopt a multimodal vaccine program to increase their patients' vaccine rates.
  Interventions: Behavioral: Multimodal Vaccine Program
- Control Practices (No Intervention): Control offices will offer usual health care related to immunizations throughout the duration of the study.

INTERVENTIONS:
Behavioral: Multimodal Vaccine Program — Efforts will be made to collaborate with private ob/gyn offices to develop a multimodal intervention to improve patients'immunization rates. As part of the overall intervention, intervention practices will agree to 1) purchase, stock, and administer influenza, HPV, and Tdap vaccines, if not already doing so and 2) track patients' vaccination status. In addition, intervention strategies adopted by intervention settings to improve immunization rates may include:
  * Patient education regarding the importance of vaccination, including encouragement of vaccination for family members
  * Practice-based reminder/recall
  * Seek to decrease missed opportunities for immunization by using either or both of the following: provider prompts and/or provider education and feedback
  Arms: Intervention Practices

SUMMARY:
The purpose of this study is to determine if a multimodal immunization program carried out in obstetrics and gynecology (ob/gyn) practices would be more effective in improving ob/gyn patients' immunization rates, specifically for Tdap (Tetanus, Diphtheria, Pertussis), HPV (Human papilloma virus), and influenza vaccines, than the usual care provided to patients in ob/gyn practices.

ELIGIBILITY:
Inclusion Criteria:

1. 15 years of age or older when presenting for care
2. Patients who present for care one year prior to the start of the intervention and up to 21 months after the start of the intervention

Exclusion Criteria:

1. less than 15 years of age when presenting for care
2. patient is not eligible for any immunizations

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97087 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in the percent of women vaccinated with one or more Tdap vaccines (among eligible patients) in intervention settings compared to control settings. | 1 year (administrative data) & 2 months (survey data) prior to intervention & 12 and 21 months after intervention (administrative and survey data)
  The percent of eligible patients presenting for care who receive Tdap vaccine will be assessed one year prior to the intervention and 12 and 21 months after the intervention. This assessment will occur in both intervention and control settings using two data sources 1) administrative data and 2) patient self-report of vaccine history.
Change in the percent of women vaccinated with influenza vaccine (among eligible patients) in intervention settings compared to control settings. | 1 year (administrative data) & 2 months (survey data) prior to intervention & 12 and 21 months after intervention (administrative and survey data)
  The percent of eligible patients presenting for care who receive influenza vaccine will be assessed one year prior to the intervention and at 12 and 21 months after the intervention. This will be assessed in both intervention and control settings using two data sources 1) administrative data and 2) patient self-report of vaccine history.
Change in the percent of women who have initiated the HPV vaccine series (among eligible patients) in intervention settings compared to control settings. | 1 year (administrative data) & 2 months (survey data) prior to intervention & 12 and 21 months after intervention (administrative and survey data)
  The percent of eligible patients presenting for care who have received one or more HPV vaccines will be assessed one year prior to the intervention and at 12 and 21 months after the intervention. This number will be assess in both intervention and control settings using two data sources 1) administrative data and 2) patient self-report of vaccine history.
Change in the percent of women who have received one or more needed vaccines (eligible patients who receive HPV, influenza, and/or Tdap vaccines) in intervention settings compared to control settings. | 1 year (administrative data) & 2 months (survey data) prior to intervention & at 12 and 21 months after intervention (administrative and survey data)
  The percent of eligible patients presenting for care who have received one or more needed vaccines (HPV, Tdap, and/or influenza vaccines) will be assessed one year prior to the intervention and at 12 and 21 months after the intervention. This number will be assess in both intervention and control settings using two data sources 1) administrative data and 2) patient self-report of vaccine history.

SECONDARY OUTCOMES:
Change in the percent of women who have completed the HPV vaccine series (among eligible patients) in intervention settings compared to control settings. | 1 year (administrative data) & 2 months (survey data) prior to intervention & at 12 and 21 months after intervention (administrative and survey data)
  The percent of eligible patients presenting for care who have completed the HPV vaccine series will be assessed one year prior to the intervention and at 12 and 21 months after the intervention. This number will be assess for both intervention and control settings using two data sources 1) administrative data and 2) patient self-report of vaccine history.
Change in the percent of women who report Tdap vaccine uptake among individuals in frequent contact with their infant in intervention offices compared to control offices | Feb/March 2013 & Feb/March 2014
  The percent of patients who report one or more individuals who are/will be in frequent contact with their infant having received Tdap vaccine will be assessed during Feb/March 2013 and Feb/March 2014. These data will be collected in patients of both intervention and control settings via on-line survey and be administered to patients who volunteer to take the survey.
Change in the percent of women who report influenza vaccine uptake among individuals in frequent contact with their infant in intervention offices. compared to control offices | Feb/March 2013 & Feb/March 2014
  The percent of patients who report one or more individuals who are/will be in frequent contact with their infant having received influenza vaccine will be assessed during Feb/March 2013 and Feb/March 2014. These data will be collected in patients of both intervention and control settings via on-line survey and be administered to patients who volunteer to take the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado Denver, Children's Hospital Colorado; Amanda Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Children's Hospital Colorado
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] O'Leary ST, Pyrzanowski J, Brewer SE, Sevick C, Miriam Dickinson L, Dempsey AF. Effectiveness of a multimodal intervention to increase vaccination in obstetrics/gynecology settings. Vaccine. 2019 Jun 6;37(26):3409-3418. doi: 10.1016/j.vaccine.2019.05.034. Epub 2019 May 15. PMID 31103367